CLINICAL TRIAL: NCT05571410
Title: Program Design Hypertension Chat Bot Pilot Study With the Primary Care Service Line
Brief Title: BP PAL - Hypertension Chat Bot Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 852102
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
Keywords: remote monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients assigned to intervention arm will a text message notifying them of enrollment, be mailed a BP cuff and receive a recruitment phone call if nonresponsive to text. If the patient does not opt out, the research coordinator will mail a blood pressure cuff and proper measurement instructions and start their remote monitoring program in the Way to Health platform. Intervention arm participants will also receive usual care. Usual care for hypertension is as needed determined by the clinical expertise of the primary care provider and can include regular follow-up visits (in person or virtual), home blood pressure readings, titration of medications during visits or via telephone, referral to specialty care (e.g., Nephrology or Cardiology), blood tests or imaging studies.
  Interventions: Behavioral: HTN Chat bot
- Control (No Intervention): Patients in the usual care arm will not be contacted by study staff at the start of the pilot, they will not receive a blood pressure cuff, and they will not receive any text messaging or any component of the program. They will eventually be contacted by study staff to schedule the 6 month BP check. Usual care for hypertension is as needed determined by the clinical expertise of the primary care provider and can include regular follow-up visits (in person or virtual), home blood pressure readings, titration of medications during visits or via telephone, referral to specialty care (e.g., Nephrology or Cardiology), blood tests or imaging studies.

INTERVENTIONS:
Behavioral: HTN Chat bot — Remote monitoring via automated messaging program
  Arms: Intervention

SUMMARY:
A 2-arm randomized pilot trial aimed at evaluating the effectiveness of a 6-month remote monitoring program for the management of hypertension (HTN). 300 eligible patients will be randomized in a 1:1 ratio into two recruitment arms: A) Control (usual care), or B) Remote monitoring via automated messaging program. The target population are patients at the Penn Family Medicine University City and Westtown primary care practices with baseline poor blood pressure control as indicated by two blood pressures greater than 140/90 within the past twelve month including the most recent measurement and on at least one anti-hypertensive agent.

DETAILED DESCRIPTION:
STUDY DESIGN:

Pragmatic, non-blinded, randomized controlled trial.

Randomization and enrollment:

* Randomization will be at the patient level (stratified/balanced randomization by PCP)
* Enrollment will take place over short time period based off of lists of eligible patients pulled from the EMR
* Lists of eligible patients sent to PCPs with opportunity to opt patients out. Patients will be contacted via text followed by phone call to introduce them to the program.

We expect recruitment to take approximately 1 month to reach a target sample size of 300. The program itself will be 6 months from the date of randomization. Total study duration should be approximately 7 months. Data analyses will take an additional 3 months.

The control group will receive usual care as determined by PCP (control arm will not receive BP cuffs).The Intervention Group will receive the BP cuff and weekly SMS messages asking for the BP reading. The methods section below will outline the details for both groups.

ELIGIBILITY:
Inclusion Criteria:

* 1) Two blood pressures > 140/90 within the past 12 months, including the most recent measurement AND 2) On at least one anti-hypertensive agent AND 3) On HTN registry AND 4)On PCSL registry 5) Are active patients at the Penn Family Medicine University City, Penn Presby and Westtown practices

Exclusion Criteria:

* Any patients meeting the following criteria are excluded from the study:

  * On a PCSK9 inhibitor medication
  * Pregnant or currently breastfeeding
  * Have a significant disability or markedly shortened life expectancy (metastatic cancer, on hospice, ESRD, dementia, end stage renal failure, congestive heart failure)
  * Not fluent in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | six months
  change in systolic blood pressure from baseline to 6 month visit

SECONDARY OUTCOMES:
Diastolic Blood Pressure | six months
  comparison of diastolic blood pressure in the control arm and intervention arm at 6 month study visit

CONTACTS AND LOCATIONS:
Overall Officials: Anna U Morgan, M.D., Principal Investigator — University of Pennsylvania; Eric Bressman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bressman E, Profka K, Norton L, Clark K, Mahraj K, Walker Z, Reid-Bey L, Girard A, Rareshide C, Xu L, Zhu J, Putt M, Volpp KG, Morgan AU. Automated Text Message-Based Program to Improve Uncontrolled Blood Pressure in Primary Care Patients: A Randomized Clinical Trial. J Gen Intern Med. 2025 May;40(6):1248-1254. doi: 10.1007/s11606-024-09225-4. Epub 2024 Dec 4. PMID 39633105